CLINICAL TRIAL: NCT06172062
Title: Establishment and Application of an Artificial Intelligence Algorithm for Automatic Identification of Intraoperative Bleeding During Laparoscopic Pancreaticoduodenectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinrui Zhu，MD (Other)
Responsible Party: Sponsor-Investigator, Xinrui Zhu，MD, attending doctor, West China Hospital
Organization: West China Hospital (Other)
Other Study IDs: 2023-1663-2
Record Dates: First submitted 2023-11-08; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Laparoscopic Pancreaticoduodenectomy
Keywords: laparoscopic pancreaticoduodenectomy; surgical videos; artificial intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LPD cohort: surgical videos of laparoscopic pancreaticoduodenectomy with label to build and test the algorithms.
  Interventions: Other: laparoscopic pancreaticoduodenectomy

INTERVENTIONS:
Other: laparoscopic pancreaticoduodenectomy — we recorded the surgical videos of laparoscopic pancreaticoduodenectomy, and labeled the information in the video to build and test the algorithms.

SUMMARY:
Surgeons will label surgical videos of laparoscopic pancreaticoduodenectomy with bleeding information from multicenter. The labeled surgical video will be used as training material to train the algorithmic model so as to build an artificial intelligence algorithm that can automatically identify intraoperative bleeding in this surgery. Then, we will test the performance capability of the algorithm.

ELIGIBILITY:
Inclusion Criteria:

1. surgical videos that recorded complete laparoscopic pancreaticoduodenectomy including resection and reconstruction phases.

Exclusion Criteria:

1.surgical videos that recorded laparoscopic pancreaticoduodenectomy combined with resection and reconstruction of mesentericoportal vein.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients underwent laparoscopic pancreaticoduodenectomy for benign and malignant diseases. Besides, the surgical videos had been recorded.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
performance of artifical intelligence algorithm | through study completion, an average of 1 month
  test the performance of the algorithm , including accuracy

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No